CLINICAL TRIAL: NCT01518920
Title: A Double-Blind, Randomized, Placebo-Controlled, Single-Dose, Crossover Study Of The Safety And Efficacy Of Two Fixed Doses Of PF-04958242 In Subjects With Age-Related Sensorineural Hearing Loss
Brief Title: A Study Of The Effects Of PF-04958242 In Subjects With Age-Related Hearing Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B1701005
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Age related sensorineural hearing loss; PF-04958242
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04958242 (Experimental)
  Interventions: Drug: PF-04958242
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04958242 — PF-04958242 0.35 mg oral solution
  Arms: PF-04958242
Drug: PF-04958242 — PF-04958242 0.27 mg oral solution
  Arms: PF-04958242
Drug: Placebo — Placebo oral solution
  Arms: Placebo

SUMMARY:
The objective of this study is to examine the safety, tolerability, and effects on hearing thresholds of two single doses of PF-04958242 and placebo in subjects with age-related hearing loss.

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a current diagnosis of age related sensorineural hearing loss in the range of 30-60 dB, averaged over 2 and 4 kHz in at least one ear.
* Subjects must have symmetric hearing loss
* Subjects who can read, speak and comprehend English.

Exclusion Criteria:

* Subjects who have a history of sudden hearing loss and history or diagnosis of rapidly progressive idiopathic hearing loss
* Subjects who have hearing disorders other than age related sensorineural hearing loss
* Subjects with moderate or greater tinnitus
* Pregnant females; breastfeeding females; females of childbearing potential

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 1 hour post-dose in pure tone audiometry averaged over 2 and 4 kHz | 1 hour

SECONDARY OUTCOMES:
Change from baseline to 5 hours post-dose in pure tone audiometry averaged over 2 and 4 kHz | 5 hours
Change from baseline to 1 hr and 5 hrs post-dose in Speech Discrimination Score | 1 hour, 5 hours
Change from baseline to 1 hr and 5 hrs post dose in Speech In Noise Testing | 1 hour, 5 hours
Change from baseline to 1 hr and 5 hrs post dose in Tinnitus Severity Ranking Scale | 1 hour, 5 hours
Plasma PF 04958242 concentrations at 45 min post dose and following endpoint assessments at 1 and 5 hrs post dose. | 45 min, 1 hour, 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- United States (5):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- [Derived] Bednar MM, DeMartinis N, Banerjee A, Bowditch S, Gaudreault F, Zumpano L, Lin FR. The Safety and Efficacy of PF-04958242 in Age-Related Sensorineural Hearing Loss: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2015 Jul;141(7):607-13. doi: 10.1001/jamaoto.2015.0791. PMID 25997115
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1701005&StudyName=A%20Study%20Of%20The%20Effects%20Of%20PF-04958242%20In%20Subjects%20With%20Age-Related%20Hearing%20Loss